CLINICAL TRIAL: NCT00290966
Title: Open Label, Randomized Multicentre Phase II/III Study of Docetaxel in Combination With Cisplatin (CDDP) or Docetaxel in Combination With 5-Fluorouracil (5-FU) and CDDP Compared to the Combination of CDDP and 5-FU in Patients With Metastatic or Locally Recurrent Gastric Cancer Previously Untreated With Chemotherapy for Advanced Disease
Brief Title: Randomized Multicenter Study Comparing Docetaxel Plus Cisplatin and 5-FU to Cisplatin Plus 5-FU in Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6044; XRP6976E-325
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Stomach Neoplasm
Keywords: docetaxel; stomach neoplasm
MeSH Terms: conditions — Stomach Neoplasms

INTERVENTIONS:
Drug: XRP6976

SUMMARY:
Phase II:

Primary objective: to select one of the 2 test arms (docetaxel with cisplatin, docetaxel with cisplatin and 5-FU), based primarily on complete responses, to advance to a phase III survival comparison against the CDDP + 5-FU control arm.

Secondary objective: to evaluate the quantitative and qualitative safety profile of the 2 test groups.

Phase III:

Primary objective: to detect a statistically significant increase in time to progression (TTP) for the test arm (docetaxel plus cisplatin and 5-FU) relative to the control arm (cisplatin plus 5-FU).

Main secondary objective: to detect a statistically significant increase in overall survival (OS) for the test arm (docetaxel plus cisplatin and 5-FU) relative to the control arm (cisplatin plus 5-FU).

Other secondary objectives: to compare response rates, time to treatment failure, duration of response, safety profiles, quality of life and disease-related symptoms.Socio-economic data will be collected in order to be able to perform an analysis by country when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient's consent form obtained, signed and dated before beginning specific protocol procedures.
* Gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction, histologically proven.
* Measurable and/or evaluable metastatic disease; if a single metastatic lesion is the only manifestation of the disease, cytology or histology is mandatory. Locally recurrent disease is accepted provided that there is at least one measurable lesion (e.g. lymph node).
* Performance status Karnofsky index > 70%.
* Life expectancy of more than 3 months.
* Adequate haematological and biochemistry parameters
* No prior palliative chemotherapy, previous adjuvant (and/or neo-adjuvant) chemotherapy is allowed if more than 12 months has elapsed between the end of adjuvant (or neo-adjuvant) therapy and first relapse.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measures.
* Other tumor type than adenocarcinoma (leiomyosarcoma ; lymphoma).
* Any prior palliative chemotherapy. Prior adjuvant (and/or neo-adjuvant) chemotherapy with a first relapse within 12 months from the end of adjuvant (or neo-adjuvant).
* Prior treatment with taxanes. Prior CDDP as adjuvant (and/or neo-adjuvant) chemotherapy with cumulative dose > 300 mg/m².

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610
Dates: Start 1998-10; Study Completion 2003-05

PRIMARY OUTCOMES:
to detect a significant increase in time to progression in favor of docetaxel plus cisplatin and 5-FU compared to cisplatin plus 5-FU. Tumor assessments (assessed with WHO criteria) had to be performed every 8 weeks until progression

SECONDARY OUTCOMES:
Patients were to be followed until death (overall survival). Clinical and laboratory were assessed with NCIC-CTG scale, before each cycle. Quality of life and clinical benefit were assessed every 2 weeks until progression and then every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Texas, US; E. Van Cutsem, MD, Principal Investigator — University hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Result] Van Cutsem E, Moiseyenko VM, Tjulandin S, Majlis A, Constenla M, Boni C, Rodrigues A, Fodor M, Chao Y, Voznyi E, Risse ML, Ajani JA; V325 Study Group. Phase III study of docetaxel and cisplatin plus fluorouracil compared with cisplatin and fluorouracil as first-line therapy for advanced gastric cancer: a report of the V325 Study Group. J Clin Oncol. 2006 Nov 1;24(31):4991-7. doi: 10.1200/JCO.2006.06.8429. PMID 17075117